CLINICAL TRIAL: NCT02698657
Title: A Phase 1, Randomized, Placebo-controlled, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASP5094 Following Multiple Intravenous Doses in Subjects With Rheumatoid Arthritis on Methotrexate
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASP5094 Following Multiple Intravenous Doses in Subjects With Rheumatoid Arthritis on Methotrexate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 5094-CL-0102; 2015-004562-28 (EudraCT Number)
Record Dates: First submitted 2016-02-10; First posted 2016-03-04 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid arthritis (RA); Methotrexate; ASP5094
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASP5094 Dose Escalation (Experimental): Three sequential cohorts will receive increasing intravenous doses of ASP5094. After all subjects in a cohort have completed study procedures the overall safety and tolerability of the dose will be determined after evaluation of the safety data. If there are no events which meet the stopping criteria, the next sequential cohort will begin enrollment while the current subjects continue through the third dose and the remainder of the study.
  Interventions: Drug: ASP5094
- Placebo Dose Escalation (Placebo Comparator): Three sequential cohorts will receive increasing intravenous doses of Placebo. After all subjects in a cohort have completed study procedures the overall safety and tolerability of the dose will be determined after evaluation of the safety data. If there are no events which meet the stopping criteria, the next sequential cohort will begin enrollment while the current subjects continue through the third dose and the remainder of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP5094 — Intravenous (IV)
  Arms: ASP5094 Dose Escalation
Drug: Placebo — Intravenous (IV)
  Arms: Placebo Dose Escalation

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of multiple ascending intravenous doses of ASP5094 in male and female subjects with rheumatoid arthritis (RA) on methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) of ≤ 35 kg/m2, inclusive, and must weigh at least 50 kg at screening.
* Subject has absolute neutrophil count within normal limits at screening. The assessment may be repeated once during screening.
* Subject has RA that was diagnosed according to the 1987 revised criteria of the American College of Rheumatology (ACR) ≥ 6 months prior to screening.
* Subject meets the ACR 1991 revised criteria for Global Functional Status in RA, Class I, II or III at screening.
* Subject MUST be on concomitant MTX:

  * for ≥ 3 months prior to day 1, and
  * at a stable dose (10 25 mg/week) for ≥ 28 days prior to day 1 and throughout the study.
* Subject's other medications taken for the treatment of RA at the time of screening must meet the noted stability requirements and remain on a stable regimen, as follows:

  * Nonsteroidal antiinflammatory drugs (NSAIDs), selective cyclooxygenase-2 (COX- 2) inhibitors, oral corticosteroids (≤ 10 mg of prednisone, or equivalent, daily) or low dose opioids (≤ 30 mg of oral morphine, or equivalent, daily) must be stable for ≥ 28 days prior to screening,
  * Hydroxychloroquine (Plaquenil®) and sulfasalazine (e.g., Azulfidine®) must have started ≥ 2 months, and be stable for ≥ 28 days, prior to day 1.
* Female subject must be either:

  * Of nonchildbearing potential: postmenopausal (defined as at least 1 year without any menses) prior to screening, or documented surgically sterile
  * Or, if of childbearing potential, Agree not to try to become pregnant during the study and for 60 days after the final study drug administration; must have a negative urine pregnancy test at screening and day 1, And, if heterosexually active, agree to consistently use 2 forms of highly effective birth control† (at least 1 of which must be a barrier method) starting at screening and throughout the study period and for 60 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 60 days.
* Female subject must not donate ova starting at screening and throughout the study period, and for 60 days after the final study drug administration.
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective forms of contraception consisting of 2 forms of birth control† (1 of which must be a barrier method) starting at screening and continue throughout the study period and for 60 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period, and for 60 days after the final study drug administration
* Subject agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Subject has an ongoing clinically significant systemic disease such as uncompensated heart failure, uncontrolled diabetes mellitus, severe hepatic failure, severe pulmonary disease or inflammatory bowel disease.
* Subject has a history of any malignancy in the past 5 years, except for adequately-treated, nonmelanoma skin cancer and adequately-treated in-situ cervical cancer.
* Subject has a history of severe allergic or anaphylactic reactions to drugs.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/ substance abuse within past 6 months prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits).
* Subject has an ongoing infection or has had an infection requiring intravenous antibiotics within 1 month prior to day 1.
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) antibody.
* Subject has a past history of serious opportunistic infection.
* Subject has a positive QuantiFERON-TB Gold test within 90 days of, or at screening, and has not completed an adequate course of antimicrobial therapy per Centers for Disease Control or local guidelines.
* Subject's laboratory test results at screening or prior to study drug dosing on day 1:

  * Outside the normal limits and considered by the investigator to be clinically significant with regard to the remaining per-protocol laboratory tests, and/or
  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) are > 2 times the upper limit of normal.
* Subject received any live or live-attenuated vaccine within 30 days prior to day 1.
* Subject received any of the following:

  * Oral or injectable gold, azathioprine, penicillamine, cyclosporine, tacrolimus or tofacitinib (Xeljanz®) within 30 days prior to day 1.
  * Anakinra (Kineret®), etanercept (Enbrel®), adalimumab (Humira®), tocilizumab (Actemra®), infliximab (Remicade®), or golimumab (Simponi®) within 60 days prior to day 1.
  * Leflunomide (Arava®) within 60 days prior to day 1, unless the subject has undergone cholestyramine washout at least 30 days prior to day 1.
  * Certolizumab (Cimzia®) and abatacept (Orencia®) within 90 days prior to day 1.
  * Rituximab (Rituxan®) or any other antiCD20 antibody, and cyclophosphamide within 180 days prior to day 1.
  * Treatment with any other conventional disease modifying antirheumatic drugs (DMARDs), or treatment with any other biologics not previously noted within 28 days or 5 half-lives, whichever is longer, prior to day 1.
* Subject has participated in a previous clinical study with treatment with ASP5094 or has participated in another dose cohort of the current trial.
* Subject has previously received an experimental agent within 28 days or 5 half-lives, whichever is longer, prior to day 1.
* Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day 1.
* Subject had surgery or has a planned elective surgery (including oral surgery) within 1 month prior to screening and 3 months after last study drug administration.
* Subject has a wound that is currently healing.
* Subject has any other condition, which in the opinion of the investigator, precludes the subject's participation in the trial.
* Subject is an employee of the Astellas group or vendors involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events | From first dose of study drug up to end of study (up to 141 days)
  A treatment-emergent adverse event (TEAE) is defined as a newly occurring or worsening adverse event (AE) observed after starting administration of study drug up until the end of study visit, inclusive. This includes abnormal laboratory tests, vital signs or electrocardiogram data that are defined as AEs if the abnormality induces clinical signs or symptoms, requires active intervention, interruption or discontinuation of study drug or is clinically significant in the investigator's opinion. A serious AE (SAE) is defined as an AE with an outcome that results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly, or birth defect or requires inpatient hospitalization or leads to prolongation of hospitalization.
Change from Baseline in Total Lymphocyte Counts | Baseline and days 29, 57, 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD19 | Baseline and days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD19/Lymphocytes | Baseline and days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD3 | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD3/Lymphocytes | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD4 | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD4/Lymphocytes | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD8 | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: CD8/Lymphocytes | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: Granulocytes | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: Granulocytes/Leukocytes | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: Natural Killer Cell Subset/Lymphocytes | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Change from Baseline in Peripheral Lymphocyte Subsets: Natural Killer Cells | Baseline and Days 29 (predose), 57 (predose), 85, 113, 141
Number of Participants with Anti-ASP5094 Antibody Formation | Days 1 (predose), 29 (predose), 57 (predose), 71, 85, 113 and 141
Area under the concentration-time curve from the time of dosing on day 1 to the end of the 4-week dosing interval for ASP5094 (AUC) | Day 1 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose
Maximum Concentration (Cmax) of ASP5094 | Day 1 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose
Time to maximum concentration (tmax) of ASP5094 | Day 1 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose
Concentration immediately prior to dosing at multiple dosing (Ctrough) for ASP5094 | Predose on days 29, 57, and 85
Accumulation ratio calculated using the maximum concentration (R3ac[Cmax]) for ASP5094 | Day 57 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose
Accumulation ratio calculated using the area under the concentration-time curve (R3ac[AUC]) for ASP5094 | Day 57 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose

SECONDARY OUTCOMES:
Terminal elimination half-life (t1/2) | Day 1 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose
Total clearance after intravenous dosing (CL) | Day 1 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose
Volume of distribution after intravenous dosing during the terminal elimination phase (VzF) | Day 1 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose
Percentage of Fluctuation | Day 1 predose, 0.5, 24, 96, 168, 216, 336, 504, 672 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (13):
- United States (7):
  - Site US10002, Anniston, Alabama
  - Site US10008, DeBary, Florida
  - Site US10004, Jacksonville, Florida
  - Site US10009, Miami Lakes, Florida
  - Site US10003, Duncansville, Pennsylvania
  - Site US10010, Memphis, Tennessee
  - Site US10001, Dallas, Texas
- Poland (6):
  - Site PL48009, Elblag
  - Site PL48011, Krakow
  - Site PL48006, Lodz
  - Site PL48007, Stalowa Wola
  - Site PL48003, Warsaw
  - Site PL48008, Wroclaw

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=326